CLINICAL TRIAL: NCT01298011
Title: A Pilot Phase II Multi Center Study of Gemcitabine and Nab-paclitaxel (Abraxane) as Preoperative Therapy for Potentially Operable Pancreatic Cancer
Brief Title: Study of Gemcitabine and Abraxane to Treat Potentially Operable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pancreatic Cancer Research Team (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCRT 10-001
Record Dates: First submitted 2011-02-14; First posted 2011-02-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Resectable Pancreatic Cancer
Keywords: operable; pancreas; Abraxane; Gemcitabine; Preoperative; potentially; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine & Abraxane Pancreatic Cancer (Experimental)
  Interventions: Drug: Gemcitabine and Abraxane

INTERVENTIONS:
Drug: Gemcitabine and Abraxane — 3 treatments for gemcitabine and abraxane every 28-days for 3 months, prior to surgery.
  Other Names: nab-paclitaxel; gemzar

SUMMARY:
The main purpose of this research study is to evaluate whether Abraxane and gemcitabine are effective in treating patients with operable pancreatic cancer.

DETAILED DESCRIPTION:
The best outcome for a patient diagnosed with pancreatic cancer is surgery. However many patients have recurrence of the cancer after successful surgery. The investigators are evaluating chemotherapy before surgery, which is a new approach.

In this study, Abraxane and gemcitabine will be tested as treatment for people with operable pancreatic cancer to see if surgery can be successfully performed and if treatment will reduce cancer cells in the tumor at surgery.

Abraxane is approved by the US FDA for the treatment of metastatic breast cancer after failure of combination chemotherapy for metastatic disease or relapse within 6 months of adjuvant chemotherapy. Gemcitabine is approved by the FDA for first line treatment for patients with locally advanced or metastatic cancer of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically or cytologically confirmed potentially resectable adenocarcinoma of the pancreas. Patients with islet cell neoplasms are excluded.

   Definition of potentially operable disease
   1. Staging by high-quality, pancreatic protocol, helical abdominal computed tomography required (Endoscopic ultrasound is not required).
   2. No extension to superior mesenteric artery (SMA) and hepatic artery.
   3. Clear fat plane between the SMA and celiac axis.
   4. No extension to celiac axis and hepatic artery.
   5. Patent superior mesenteric vein and portal vein.
   6. No evidence of distant or extra-hepatic disease by CT scans.
   7. Pretreatment histological or cytological confirmation of an adenocarcinoma.
2. Male or non-pregnant and non-lactating female, and ≥ 18 years of age.
3. If a female patient is of child-bearing potential, she must have a negative serum pregnancy test (β hCG) documented within 72 hours of the first administration of study drug.
4. If sexually active, the patient must agree to use contraception considered adequate and appropriate by the Investigator.
5. Patient must have received no prior chemotherapy or radiation for pancreatic cancer and no exposure to gemcitabine and/or Abraxane
6. Patient has the following blood counts at baseline:

   1. ANC ≥ 1.5 x 109/L (1500 /mm³);
   2. Platelets ≥ 100 x 109/L; (100,000/mm³);
   3. Hgb ≥ 10 g/dL.
7. Patient has the following blood chemistry levels at baseline:

   1. AST (SGOT), ALT (SGPT) ≤ 2.5 x upper limit of normal (ULN);
   2. Alkaline phosphatase (AP) ≤ 2.5 X ULN;
   3. Total bilirubin ≤1.5 mg/dl;
   4. Serum creatinine ≤1.5mg/dl or calculated clearance ≥ 50 mL/min/1.73 m² for patients with serum creatinine levels >1.5 mg/dl.
8. Patient has acceptable coagulation status as indicated by a PT within normal limits (±15%) and PTT within normal limits (± 15%).
9. Patient has an ECOG performance status PS 0-1.
10. Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form prior to participation in any study-related activities.

Exclusion Criteria:

1. Patient has borderline resectable disease
2. Patient uses therapeutic coumadin for a history of pulmonary emboli or DVT.
3. Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
4. Patient has known infection with HIV, hepatitis B, or hepatitis C.
5. Patient has undergone major surgery, other than diagnostic surgery (i.e.--surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
6. Prior chemotherapy or radiation for pancreatic cancer. Prior exposure to gemcitabine and/or Abraxane.
7. Patient has a history of allergy or hypersensitivity to the study drugs.
8. Patient has serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the patient to receive an experimental research drug.
9. Patient is unwilling or unable to comply with study procedures.
10. Patient is enrolled in any other therapeutic clinical protocol or investigational trial.
11. Patient has metastatic disease on radiological staging.
12. Patients aged ≥ 80 are not excluded. As two events of fatal sepsis have been seen in this group in other studies, candidates in this age group should be thoroughly evaluated before enrollment in the study, to ensure they are fit to receive chemotherapy. In addition to meeting all of the baseline patient selection criteria, clinical judgment on their susceptibility to infection and expected stability of their performance status as to receive repeat weekly chemotherapy cycles, should be paid special attention to. Patients should not be enrolled in the study should there be any hesitation on any of these considerations. Baseline criteria for all patients enrolled on the study must be carefully evaluated and all criteria followed appropriately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Grade III/IV histological response in tumor specimen rate after induction therapy. | At time of surgery

SECONDARY OUTCOMES:
Number of participants with adverse events. | From the initial dose of study drug up to 28 days after last dose of study drug.
Tumor response rate to therapy. | Baseline and 16 weeks
  Pre and post therapy radiological assessments of the primary tumor will be compared using RECIST criteria.
Change in CA 19-9 | Baseline, Day 1 of each cycle, and end of therapy.
  Baseline CA19-9 and subsequent levels will be compared.
Resection rate at surgery | At time of surgery
  The number of patients who have R0 and R1 surgery will be compiled.
Time to recurrence | Time from first dose of study drug to date of first documented progression or date of death, whichever occurs first, assessed up to 60 months.
SPARC protein expression in tumor | At time of surgery
Overall Survival | Time from the first dose of study drug until date of death from any cause, up to 60 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh K. Ramanathan, MD, Principal Investigator — TGen Drug Development
Locations (4):
- United States (4):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - St Mary's / Trinity Health Care, Grand Rapids, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania